CLINICAL TRIAL: NCT00928057
Title: Comparison of Glycemic Control Among Diabetics Using the 4mm x 32G BD Pen Needle Versus the 8mm x 31G BD Pen Needle and the 5mm x 31G BD Pen Needle
Brief Title: Comparison of Glycemic Control Among Diabetics Using Three Different Pen Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Dr. Kenneth Kassler-Taub / WW Vice President / Medical Affairs, BD Medical
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BDDC-08-011
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Pen Needle; Diabetes; Insulin; Glycemic; Pain; Fructosamine; Leakage; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance; Pain; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 mm / 8 mm PN (Experimental): Subjects randomized to this study arm used either the 4mm PN or the 8mm PN for 3 weeks, then switched to the alternate PN for another 3 weeks. Order of PN use was randomly determined.
  Interventions: Device: 4mm x 32G pen needle; Device: 8mm x 31G pen needle
- 4 mm / 5 mm PN (Experimental): Subjects randomized to this study arm used either the 4mm PN or the 5mm PN for 3 weeks, then switched to the alternate PN for another 3 weeks. Order of PN use was randomly determined.
  Interventions: Device: 4mm x 32G pen needle; Device: 5mm x 31G pen needle

INTERVENTIONS:
Device: 4mm x 32G pen needle — For 3 weeks, subjects used this pen needle with their own pen device for all daily insulin injections they usually administered themselves with a pen device. Subjects followed their usual insulin regimen and there was no upper limit on total daily insulin dosage or number of injections. Subjects were advised to inject straight in when using the 4mm PN, with no pinch up.
  Other Names: BD Ultra-Fine™ Nano pen needle, Catalog number 320122
Device: 8mm x 31G pen needle — For 3 weeks, subjects used this pen needle with their own pen device for all daily insulin injections they usually administered themselves with a pen device. Subjects followed their usual insulin regimen and there was no upper limit on total daily insulin dosage or number of injections. Subjects were directed to use pinch-up when injecting in the abdomen or thigh with the 8mm PN, and no pinch-up at other injection sites.
  Other Names: BD Ultra-Fine™ Short pen needle, Catalog number 320109
  Arms: 4 mm / 8 mm PN
Device: 5mm x 31G pen needle — For 3 weeks, subjects used this pen needle with their own pen device for all daily insulin injections they usually administered themselves with a pen device. Subjects followed their usual insulin regimen and there was no upper limit on total daily insulin dosage or number of injections. Subjects were advised to inject straight in when using the 5mm PN, with no pinch up.
  Other Names: BD Ultra-Fine™ Mini pen needle, Catalog Number 320119
  Arms: 4 mm / 5 mm PN

SUMMARY:
Anxiety about needles is a commonly expressed concern by diabetics about beginning insulin therapy. A shorter, thinner pen needle that delivers insulin with the safety and efficacy profile of currently marketed pen needles may appeal to many diabetic patients as the new needle may be perceived as less intimidating and more comfortable. Currently marketed pen needles range in length from 5 to 12.7 millimeters (mm).

The primary purpose of this study was to evaluate whether the investigational 4mm x 32 Gauge(G) pen needle manufactured by Becton, Dickinson and Company (BD) provides equivalent glucose control (as measured by fructosamine levels) as the currently marketed BD 5mm x 31 G and BD 8mm x 31 G pen needles (PN)in diabetic subjects with varying insulin dosage regimens.

DETAILED DESCRIPTION:
Within each dose group, subjects were randomly assigned at baseline to one of two study arms. One study arm (4/5 mm PN) compared the BD 4mm PN to the 5mm PN, and the other arm (4/8 mm PN) compared the BD 4mm PN to the 8mm PN, in a crossover fashion. Based on the randomization, subjects used either the 4mm or the other assigned PN (5mm or 8mm) for the first 3 weeks, then switched to the alternate PN for the next 3 weeks. Glycemic control was assessed by serum fructosamine (FRU) levels at the end of each 3 week period.

Based on their baseline insulin regimen, subjects were also assigned to an insulin dosing group (Low or Regular) to help ensure balance among treatment arms. Requirements for each group were as follows: Low Dose: largest single dose of insulin each day with a pen device must be less than or equal to 20 units. Regular Dose: largest single dose of insulin each day, with a pen device, must be 21-40 units.

Explanation of Visits and Timing of Assessments:

Visit 1:

* Screening
* Informed Consent
* Demographics
* Inclusion /Exclusion
* Hemoglobin A1c measurement (HbA1c)

Visit 2 (Baseline:)

* Insulin dose group assignment (Low dose or Regular dose)
* Randomization
* Fructosamine blood sample collected
* Dispense pen needle (PN) assigned first

Visit 3 (approximately 3 weeks after starting first PN)

* Pain rated by subject relative to baseline PN
* Review Adverse Events (AEs) and reported events of injection site leakage
* Fructosamine blood sample collected
* Dispense second assigned PN

Visit 4 (approximately 3 weeks after starting second PN):

* Review AEs and reported events of injection site leakage
* Fructosamine blood sample collected
* Pain rated relative to previously used PN
* Study Completion

ELIGIBILITY:
Inclusion Criteria:

* Insulin requiring diabetics (type 1 or type 2)
* Using a pen device for injections at least once per day, for at least two months prior to baseline (Study Visit Two).
* 18 to 75 years of age, inclusive.
* Body Mass Index from 18 to 50 kg/m², inclusive.
* Hemoglobin A1c from 5.5 to 9.5 percent (%), inclusive.
* Largest single dose of insulin a day less than or equal to 40 units

Exclusion Criteria:

* Current status or history of a medical condition that would contraindicate treatment with the study product or other conditions which, in the opinion of the Investigator, would place the subject at risk or have the potential to confound interpretation of the study results (i.e. recent history of ketoacidosis, hypoglycemic unawareness, etc.).
* Hemophilia or any other disorder which causes excessive bleeding or requires frequent transfusions.
* History of intravenous drug abuse (self-reported).
* Bleeding disorder, hemophilia or subject is currently taking anti-coagulant medications (e.g., heparin, Coumadin®, warfarin).
* Self-reported blood borne infection.
* Pregnant (from medical history only).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kassler-Taub, MD, Study Director — Becton, Dickinson and Company
Locations (4):
- United States (4):
  - Radiant Research, Birmingham, Alabama
  - AMCR Institute, Inc., Escondido, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rainier Clinical Research Center, Inc., Renton, Washington

REFERENCES:
- [Result] Hirsch LJ, Gibney MA, Albanese J, Qu S, Kassler-Taub K, Klaff LJ, Bailey TS. Comparative glycemic control, safety and patient ratings for a new 4 mm x 32G insulin pen needle in adults with diabetes. Curr Med Res Opin. 2010 Jun;26(6):1531-41. doi: 10.1185/03007995.2010.482499. PMID 20429832
- [Derived] Hirsch LJ, Gibney MA, Li L, Berube J. Glycemic control, reported pain and leakage with a 4 mm x 32 G pen needle in obese and non-obese adults with diabetes: a post hoc analysis. Curr Med Res Opin. 2012 Aug;28(8):1305-11. doi: 10.1185/03007995.2012.709181. Epub 2012 Jul 18. PMID 22762347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at four independent research centers/diabetes clinics from June 2009 - October 2009
Pre-assignment Details: A total of 205 subjects were screened at four sites. Of those, 32 subjects did not satisfy eligibility criteria or withdrew consent prior to using the test products, and the remaining 173 subjects were enrolled and randomized.
Groups:
- 4 mm / 8 mm PN: This group represents all subjects that were randomized to compare the 4mm and 8mm pen needle (PN) during the study. Each PN was used for 3 consecutive weeks; which PN was used first was based on the subject's randomization assignment.
- 4 mm / 5 mm PN: This group represents all subjects that were randomized to compare the 4mm and 5mm pen needle (PN) during the study. Each PN was used for 3 consecutive weeks; which PN was used first was based on the subject's randomization assignment.
Period: Overall Study
Arm/Group | 4 mm / 8 mm PN | 4 mm / 5 mm PN
Started | 84 | 89
Completed | 82 | 85
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 4 mm / 8 mm PN: This group represents all subjects that were randomized to the study arm comparing the 4 mm and 8 mm pen needles, regardless of whether they completed the study.
- 4 mm / 5 mm PN: This group represents all subjects that were randomized to the study arm comparing the 4 mm and 5 mm pen needles, regardless of whether they completed the study.
- Total: Total of all reporting groups
Arm/Group | 4 mm / 8 mm PN | 4 mm / 5 mm PN | Total
Number analyzed (Participants) | 84 | 89 | 173
Age Continuous [Mean (Full Range); unit: years] | 51.3 [18.1 to 76.0] | 53.8 [22.3 to 76.2] | 52.6 [18.1 to 76.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 75
  Male | 48 | 50 | 98
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian | 67 | 66 | 133
  Black/African American | 10 | 16 | 26
  Hispanic/Latino | 1 | 2 | 3
  Asian | 4 | 4 | 8
  More than one race | 2 | 1 | 3
Diabetes Type [Number; unit: Participants]
  Type 1 diabetes | 30 | 34 | 64
  Type 2 diabetes | 54 | 55 | 109
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m²] | 30.1 [20 to 49] | 30.9 [21 to 48] | 30.5 [20 to 49]
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent] — A blood sample for HbA1c was collected at screening
  percent | 7.4 (1.0) | 7.6 (1.0) | 7.5 (1.0)
Insulin Dose Group [Number; unit: participants] — Subjects were assigned to an insulin dosing group (Low or Regular) based on their baseline regimen to help ensure balance among treatment arms. Low Dose: largest single dose of insulin a day, with a pen device, was <=20 units. Regular Dose: largest single dose of insulin a day, with a pen device, 21-40 units.
  participants
    Low Dose | 48 | 49 | 97
    Regular Dose | 36 | 40 | 76
Single Largest Daily Insulin Dose [Mean (Full Range); unit: Units] — At baseline, subjects described their current insulin regimen, including the largest single daily insulin dose self-administered with a pen needle.
  Units | 19.6 [2 to 40] | 21.3 [2 to 40] | 20.5 [2 to 40]
Serum Fructosamine Concentration [Mean (Standard Deviation); unit: umol/L] — A blood sample was collected at baseline (Visit 2).
  umol/L | 298.3 (48.4) | 301.5 (61.0) | 299.9 (55.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent (%) Absolute Change in Fructosamine
Description: Within each study arm (4mm / 5mm PN, or 4mm / 8mm PN) subjects used one pen needle (PN) for 3 weeks then switched to the alternate PN for the next three weeks, for a total of 6 weeks. The principal endpoint measure of glycemic control is the percent absolute change in serum fructosamine concentration, based on the fructosamine (FRU) concentration measured in micromoles per liter (umol/L) at the end of each three week period. The change was calculated according to the following formula:
  Percent absolute change in FRU, or %|∆ FRU|= 100*[FRU(4mm)-FRU(5 or 8mm)]/[FRU(5 or 8mm)].
Time Frame: 3 weeks per pen needle, from visit 2-3 and visit 3-4.
Population: 167 subjects completed the study. 163 of the 167 completed subjects were included in this analysis. Four (4) of 167 were excluded due to out of window fructosamine samples (3), or laboratory error with fructosamine sample (1).
Measure: Mean (95% Confidence Interval); unit: Percent absolute change
Groups:
- 4 mm / 8 mm PN; 4 mm / 5 mm PN: use of one PN for insulin injections for 3 weeks, followed by 3 weeks with the alternate PN
Arm/Group | 4 mm / 8 mm PN | 4 mm / 5 mm PN
Number analyzed (Participants) | 80 | 83
Percent absolute change | 5.5 [4.5 to 6.4] | 4.9 [3.8 to 6.0]
Statistical Analysis 1: Comparison: 4 mm / 8 mm PN; The effects of pen needle type on glycemic control were tested for statistical significance using analysis of variance (ANOVA). The ANOVA model was used to calculate the absolute percent (%)change in fructosamine (% |∆ Fru|), with 95 % confidence intervals; Test type: Non-Inferiority or Equivalence — To conclude equivalence for glycemic control, the average absolute percent change in fructosamine and 95% confidence interval had to be within 20%. 80 subjects were required to be in each insulin dose group (40 per PN arm) to provide 90% power for an equivalence with alpha=0.05; p = 0.506, ANOVA — The threshold for statistical significance, or alpha, is 0.05; The ANOVA model has effects for subject, insulin dose group, investigator site and order of pen needle use
Statistical Analysis 2: Comparison: 4 mm / 5 mm PN; The effects of pen needle type on glycemic control were tested for statistical significance using ANOVA. The ANOVA model was used to calculate the % |∆ Fru|, with 95% confidence intervals; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.878, ANOVA — The threshold for significance, or alpha, is 0.05; The ANOVA model has effects for subject, insulin dose group, investigator site and order of pen needle use

2. Secondary Outcome: Percent Absolute Change in Fructosamine, by Dose Group
Description: Glycemic control was determined separately for each insulin dose group in the same manner as described for the primary outcome measure, according to the following formula:
  %|∆ FRU|= 100*[FRU(4mm)-FRU(5 or 8mm)]/[FRU(5 or 8mm)].
Time Frame: 3 weeks per pen needle, from visit 2-3 and visit 3-4.
Population: 4 of the 167 completed subjects were excluded for out of window fructosamine samples (3), or lab error with a sample (1).
  For 4 mm/8 mm: this includes 45 subjects in the Low Dose insulin group and 35 in the Regular Dose group. For 4 mm/5 mm: this includes 47 subjects in the Low Dose insulin group and 36 in the Regular Dose group.
Measure: Mean (95% Confidence Interval); unit: Percent absolute change
Arm/Group | 4 mm / 8 mm PN | 4 mm / 5 mm PN
Number analyzed (Participants) | 80 | 83
Percent absolute change
  Low Insulin Dose Group | 5.5 [4.4 to 6.7] | 5.5 [3.7 to 7.2]
  Regular Insulin Dose Group | 5.3 [3.7 to 7.0] | 4.2 [3.0 to 5.3]

3. Secondary Outcome: Number of Subjects With Severe Unexplained Hypoglycemic Events
Description: Severe Unexplained Hypoglycemia is defined as an event in which the subject's blood glucose is below 50 milligrams per deciliter (mg/dL) and/or they required assistance from another person for treatment and there is no identified cause (for example, the subject skipped a meal). These events were also reported as Adverse Events.
Time Frame: During 3 weeks using each pen needle
Population: All subjects that were randomized and used at least one of the study pen needles are included. The number of subjects with one or more events while using each PN is presented.
Measure: Number; unit: participants
Groups:
- 4 mm PN: All randomized subjects that used the 4mm PN, either during the first or second 3 weeks of the study.
- 5 mm PN: All randomized subjects that used the 5mm PN, either during the first or second 3 weeks of the study.
- 8 mm PN: All randomized subjects that used the 8mm PN, either during the first or second 3 weeks of the study.
Arm/Group | 4 mm PN | 5 mm PN | 8 mm PN
Number analyzed (Participants) | 173 | 89 | 84
participants | 5 | 5 | 4

4. Secondary Outcome: Number of Subjects With Severe Unexplained Hyperglycemic Events
Description: Severe Unexplained Hyperglycemia is defined as requiring a visit to the emergency room or hospitalization and/or having a blood glucose value above 450mg/dL without an identified cause (for example, the subject missed an insulin dose). These events were also reported as Adverse Events.
Time Frame: During 3 weeks using each pen needle
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | 4 mm PN | 5 mm PN | 8 mm PN
Number analyzed (Participants) | 173 | 89 | 84
participants | 0 | 2 | 1

5. Other Pre Specified Outcome: Percentage of Subjects With at Least One Leakage Event
Description: After each insulin injection with a study pen needle, subjects recorded in their study diary if they observed insulin leakage from the injection site. Subjects were not required to make a diary entry if there was no leakage.
Time Frame: each PN was used for 3 weeks
Measure: Number; unit: percent of subjects
Groups:
- 4 mm PN: All randomized subjects that used the 4mm PN
- 5 mm PN: All randomized subjects that used the 5mm PN
- 8 mm PN: All randomized subjects that used the 8mm PN
Arm/Group | 4 mm PN | 5 mm PN | 8 mm PN
Number analyzed (Participants) | 164 | 83 | 81
percent of subjects | 44 | 47 | 56

6. Secondary Outcome: Relative Injection Pain Score Assessed by Subject
Description: After using the second assigned pen needle (PN) for 3 weeks, subjects used a 150mm Visual Analog Scale (VAS) to rate the pain of the second PN relative to the first PN. The VAS was anchored at the center (0mm) with "as painful", and at the extreme ends with "much less painful" (-75mm) and "much more painful" (+75mm). VAS scores were adjusted for the order of PN use, such that a positive score means that the 4mm PN was scored as more painful than the reference PN (5mm or 8mm), and a negative score indicates that the 4mm PN was less painful than the reference.
Time Frame: Visit 4: 18-24 days after starting 2nd pen needle
Population: Of the 167 subjects that completed the study, 137 subjects had within-window VAS pain scores for Visit 4 and were included in this analysis. Per the protocol, the allowable visit window was 18-24 days from Visit 3, when the subject switched from the 1st to 2nd assigned pen needle.
Measure: Mean (Standard Error); unit: mm
Arm/Group | 4 mm / 8 mm PN | 4 mm / 5 mm PN
Number analyzed (Participants) | 69 | 68
mm | -23.26 (4.24) | -11.91 (5.61)
Statistical Analysis 1: Comparison: 4 mm / 5 mm PN; The null hypothesis is that the pain from the 4mm is the same or greater than the pain for the reference. The alternative hypothesis is that the pain from the 4mm is less than the pain for the reference; Test type: Superiority or Other; p = 0.019, t-test, 1 sided — The threshold for statistical significance, or alpha, is 0.05
Statistical Analysis 2: Comparison: 4 mm / 8 mm PN; As described for the 4 vs. 5mm statistical analysis; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

7. Other Pre Specified Outcome: Reported Injection Site Leakage Events, by Pen Needle Type and Droplet Size
Description: If insulin leakage from the injection site was observed, subjects rated the size of the leakage droplet based on a visual scale provided in their diaries. Scores of 1+, 2+, 3+, and 4+ correspond to droplet sizes of 1, 10, 20 and 50 ul, respectively. Droplets larger than those shown on the scale were scored as 5+. Subjects were not required to make a diary entry if there was no leakage.
Time Frame: each PN was used for 3 weeks
Population: The number of participants shown is the number of subjects that reported at least one event of leakage (see previous data table). The number of reported leakage events is presented for each droplet size category. No data were collected if there was no leakage.
Measure: Number; unit: number of events
Groups:
- 4 mm PN: Use of 4 mm PN for insulin injections for 3 weeks.
- 5 mm PN: Use of 5 mm PN for insulin injections for 3 weeks.
- 8 mm PN: Use of 8 mm PN for insulin injections for 3 weeks.
Arm/Group | 4 mm PN | 5 mm PN | 8 mm PN
Number analyzed (Participants) | 72 | 39 | 45
number of events
  1+, or 1 ul | 372 | 289 | 200
  2+, or 10 ul | 221 | 120 | 126
  3+, or 20 ul | 44 | 50 | 25
  4+, or 50 ul | 12 | 20 | 5
  5+, or > 50 ul | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: upon enrollment to study completion
Description: Adverse events collection began once subjects were enrolled and continued throughout the 6 week randomized intervention period.
  The Investigator considered all Serious Adverse Events as unlikely to be related to, or not related to, the study devices or procedures.
Groups:
- 8mm PN: All randomized subjects that used the 8 mm pen needle.
- 5mm PN: All randomized subjects that used the 5 mm pen needle.
- 4mm PN: All randomized subjects that used the 4mm pen needle.
Arm/Group | 8mm PN | 5mm PN | 4mm PN
Serious Adverse Events (participants affected / at risk) | 2/84 | 0/89 | 4/173
Other Adverse Events (participants affected / at risk) | 24/84 | 23/89 | 40/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8mm PN (N=84) | 5mm PN (N=89) | 4mm PN (N=173)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemic seizure (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Non-Hodgkins lymphoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 8mm PN (N=84) | 5mm PN (N=89) | 4mm PN (N=173)
hypoglycemia (Metabolism and nutrition disorders) | 22 | 21 | 36 — all nonserious events including severe unexplained events as defined by the protocol
hyperglycemia (Metabolism and nutrition disorders) | 4 | 7 | 7 — all nonserious events including severe unexplained events as defined by the protocol
Pain at injection site (Injury, poisoning and procedural complications) | 11 | 11 | 27 — The investigator was not required to report mild, self-limited injection site pain as an adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less